CLINICAL TRIAL: NCT01609218
Title: A Study to Evaluate the Impact of Activated Charcoal on the Absorption of LY2140023 in Healthy Subjects
Brief Title: A Study of LY2140023 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Denovo Biopharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 12858; H8Y-MC-HBCZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Results first posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2012-10

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — LY 2140023

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 80 mg LY2140023 (Experimental): Single oral dose of 80 milligrams (mg) LY2140023 administered alone
  Interventions: Drug: LY2140023
- 80 mg LY2140023 + 75 g aqueous activated charcoal (Experimental): Single oral dose of 80 mg LY2140023 followed 1 hour later by single oral dose of 75 grams (g) aqueous activated charcoal.
  Interventions: Drug: LY2140023; Drug: Aqueous activated charcoal

INTERVENTIONS:
Drug: LY2140023
Drug: Aqueous activated charcoal
  Arms: 80 mg LY2140023 + 75 g aqueous activated charcoal

SUMMARY:
The study will evaluate the effect of activated charcoal on absorption of LY2140023. The study involves a single dose of 80 milligrams (mg) LY2140023 taken as 1 tablet by mouth 2 times during study (once with activated charcoal, once without activated charcoal). This study will last approximately 16 days, not including screening. Screening is required within 28 days prior to study entry.

ELIGIBILITY:
Inclusion Criteria:

* are healthy males or females, as determined by medical history and physical examination
* male participants agree to use a reliable method of birth control during the study and for 3 months following the last dose of LY2140023, and agree not to donate sperm for 3 months following the last dose of LY2140023
* female participants:

  * of childbearing potential, who test negative for pregnancy at screening and who agree to use a reliable method of birth control during the study and for 3 months following the last dose of LY2140023
  * of non-childbearing potential; postmenopausal or permanently sterile following hysterectomy, bilateral salpingectomy or confirmed tubal occlusion (not tubal ligation). Postmenopausal is defined as spontaneous amenorrhea for at least 12 months, and a plasma follicle-stimulating hormone (FSH) level >40 milli-international units per milliliter(mIU/mL), unless the participant is taking hormone replacement therapy
* have given written informed consent approved by Lilly and the chosen ethical review board (ERB)

Exclusion Criteria:

* are currently enrolled in, have completed or discontinued within the last 90 days from, a clinical trial involving an investigational product other than the investigational product used in this study; or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* have known allergies to LY2140023 or LY404039, related compounds, activated charcoal, or any components of the formulation
* are participants who have previously withdrawn from this study or any other study investigating LY2140023 after receiving at least 1 dose of LY2140023
* show evidence or any history of significant active neuropsychiatric disease (for example, manic depressive illness, schizophrenia, depression)
* have increased risk of seizures based on a history of:

  * one or more seizures (except for a single simple febrile seizure [lacking focality and lasting less than 15 minutes, not associated with a central nervous system (CNS) infection or severe metabolic disturbance] as a child between ages 6 months to 5 years)
  * head trauma with loss of consciousness or a post-concussive syndrome within 1 year or lifetime history of head trauma with persistent neurological deficit (focal or diffuse)
  * CNS infection, uncontrolled migraine, or transient ischemic attack (TIA) within 1 year; stroke with persistent neurological deficit (focal or diffuse). Uncontrolled migraine is defined as migraine attacks that produce headache lasting up to 72 hours and are often accompanied by associated symptoms (nausea, photophobia, and phonophobia) that impair well-being and disrupt social functioning. TIA is defined as "mini-stroke" caused by temporary disturbance of blood supply to an area of the brain, which results in a sudden, brief decrease in brain function
  * CNS infection with persistent neurological deficit (focal or diffuse)
  * brain surgery
  * electroencephalogram (EEG) with paroxysmal (epileptiform) activity (isolated spikes waves, repetitive bursts of sharp waves, paroxysmal activity, frank seizures, spike-wave complexes, or sharp-slow wave complexes, or as locally defined)
  * brain structural lesion, including developmental abnormalities, as determined by examination or imaging studies (except hydrocephalus treated by shunt and without neurological deficit)
* show evidence of active renal disease (for example, diabetic renal disease, polycystic kidney disease) or creatinine clearance less than 90 milliliters per minute (mL/min) as determined by the Cockroft Gault formula
* show evidence or any history of known substance dependence or abuse at any time (according to Diagnostic and Statistical Manual of Mental Disorders [DSM-IV] diagnosis), or regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* have a clinically significant abnormality in the neurological examination
* participants judged prior to randomization to be at suicidal risk by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a 2-period crossover study. Participants received single doses of LY2140023 on 2 different occasions: 1) LY2140023 administered alone (Treatment A) and 2) LY2140023 administered and followed 1 hour later by a single dose of aqueous activated charcoal (Treatment B). Participants were randomized to Treatment Sequence AB or BA.
Groups:
- First LY2140023 Alone, Then LY2140023 + Activated Charcoal: Period 1: Single oral dose of 80 milligrams (mg) LY2140023 administered alone
  Period 2: Single oral dose of 80 mg LY2140023 followed 1 hour later by single oral dose of 75 grams (g) aqueous activated charcoal
  There was a washout period of at least 3 days between dosing occasions.
- First LY2140023 + Activated Charcoal, Then LY2140023 Alone: Period 1: Single oral dose of 80 mg LY2140023 followed 1 hour later by single oral dose of 75 g aqueous activated charcoal
  Period 2: Single oral dose of 80 mg LY2140023 administered alone
  There was a washout period of at least 3 days between dosing occasions.
Period: Period 1
Arm/Group | First LY2140023 Alone, Then LY2140023 + Activated Charcoal | First LY2140023 + Activated Charcoal, Then LY2140023 Alone
Started | 13 | 14
Received LY2140023 | 13 | 14
Received Activated Charcoal | 0 (Participants in this treatment sequence did not receive activated charcoal during Period 1.) | 12 (Two participants discontinued after receiving LY2140023 but prior to receiving activated charcoal.)
Completed | 10 | 8
Not Completed | 3 | 6
Not completed — Adverse Event | 3 | 5
Not completed — Sponsor Decision | 0 | 1
Period: Period 2
Arm/Group | First LY2140023 Alone, Then LY2140023 + Activated Charcoal | First LY2140023 + Activated Charcoal, Then LY2140023 Alone
Started | 10 | 9 (One participant did not complete Period 1 but did continue onto Period 2.)
Received LY2140023 | 10 | 9
Received Activated Charcoal | 9 | 0 (Participants in this treatment sequence did not receive activated charcoal during Period 2.)
Completed | 9 | 9
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- All Participants: This was 2-period crossover study. Participants received single oral doses of LY2140023 on 2 different occasions: 1) 80 mg LY2140023 administered alone (Treatment A) and 2) 80 mg LY2140023 administered and followed 1 hour later by a single oral dose of 75 g aqueous activated charcoal (Treatment B). Participants were randomly assigned to treatment sequence AB or BA.
Arm/Group | All Participants
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 19
Race/Ethnicity, Customized [Number; unit: participants]
  White | 24
  Black or African American | 1
  Asian | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 27

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax) of LY2140023
Description: Venous blood samples were collected for pharmacokinetic parameter estimates for LY2140023 alone and in the presence of aqueous activated charcoal.
Time Frame: Predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, and 24 hours postdose
Population: Participants who received study drug(s), did not have an incidence of vomiting following administration of LY2140023, and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- 80 mg LY2140023: Single oral dose of 80 mg LY2140023 administered alone
- 80 mg LY2140023 + 75 g Aqueous Activated Charcoal: Single oral dose of 80 mg LY2140023 followed 1 hour later by single oral dose of 75 g aqueous activated charcoal
Arm/Group | 80 mg LY2140023 | 80 mg LY2140023 + 75 g Aqueous Activated Charcoal
Number analyzed (Participants) | 18 | 14
nanograms per milliliter (ng/mL) | 251 (31) | 171 (25)

2. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-inf]) of LY2140023
Description: as for outcome 1
Time Frame: Predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, and 24 hours postdose
Population: Participants who received study drug(s), did not have an incidence of vomiting following administration of LY2140023, and had evaluable AUC(0-inf) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram hours per milliliter (ng*h/mL)
Arm/Group | 80 mg LY2140023 | 80 mg LY2140023 + 75 g Aqueous Activated Charcoal
Number analyzed (Participants) | 18 | 14
nanogram hours per milliliter (ng*h/mL) | 1120 (24) | 876 (26)

3. Primary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax) of LY404039 (Active Moiety)
Description: Venous blood samples were collected for pharmacokinetic parameter estimates for LY404039 alone and in the presence of aqueous activated charcoal.
Time Frame: Predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 80 mg LY2140023 | 80 mg LY2140023 + 75 g Aqueous Activated Charcoal
Number analyzed (Participants) | 18 | 14
ng/mL | 474 (26) | 324 (20)

4. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-inf]) of LY404039 (Active Moiety)
Description: as for outcome 3
Time Frame: Predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 9, 12, 16, and 24 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 80 mg LY2140023 | 80 mg LY2140023 + 75 g Aqueous Activated Charcoal
Number analyzed (Participants) | 18 | 14
ng*h/mL | 2780 (15) | 2190 (19)

ADVERSE EVENTS:
Arm/Group | 80 mg LY2140023 | 80 mg LY2140023 + 75 g Aqueous Activated Charcoal
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 16/22 | 13/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 80 mg LY2140023 (N=22) | 80 mg LY2140023 + 75 g Aqueous Activated Charcoal (N=24)
Nausea (Gastrointestinal disorders) | 9 (12) | 8 (8)
Vomiting (Gastrointestinal disorders) | 7 (11) | 7 (7)
Feeling hot (General disorders) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days